CLINICAL TRIAL: NCT00313911
Title: Large Scale Safety Study of a DTaP-IPV-Hep B-PRP~T Combined Vaccine, in Comparison to Tritanrix-Hep B/Hib™ and OPV Administered at 2, 4, and 6 Months of Age in Latin American Infants
Brief Title: Safety of DTaP-IPV-Hep B-PRP~T Combined Vaccine Compared to Tritanrix-HepB/Hib™ and OPV Given at Age 2, 4, and 6 Months.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A3L04
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Diphtheria; Tetanus; Pertussis; Haemophilus Influenzae Type b; Hepatitis B
Keywords: Diphtheria; Tetanus; Pertussis; Recombinant Hepatitis B; Poliomyelitis; Haemophilus influenzae type b; Tetanus protein
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Haemophilus Infections; Hepatitis B; Poliomyelitis | interventions — DTaP-IPV-HB-PRP-T vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: DTaP-IPV-Hep B-PRP-T (Experimental)
  Interventions: Biological: DTaP-IPV-HB-PRP~T
- Group 2: Tritanrix-Hep B/Hib™+OPV (Active Comparator)
  Interventions: Biological: Tritanrix-HepB/Hib

INTERVENTIONS:
Biological: DTaP-IPV-HB-PRP~T — 0.5 mL, Intramuscular (IM)
  Arms: Group 1: DTaP-IPV-Hep B-PRP-T
Biological: Tritanrix-HepB/Hib — 0.5 mL, Intramuscular
  Arms: Group 2: Tritanrix-Hep B/Hib™+OPV

SUMMARY:
To demonstrate that DTaP-IPV-HB-PRP~T combined vaccine does not induce a higher incidence rate of high fever than Tritanrix-HepB/Hib™ and Oral Polio Vaccine (OPV) after any of the three vaccinations at 2, 4, and 6 months of age for each subject.

To evaluate the overall safety in terms of:

Any solicited adverse reactions in the first 7 days after each injection, Any adverse events and reactions in the first 30 days after each injection, Any serious adverse events during the trial.

Immunogenicity:

To document the immune response to Hepatitis B antigen of the three batches of the investigational DTaP-IPV-HB-PRP~T vaccine.

ELIGIBILITY:
Inclusion Criteria:

* 2 months old infants on the day of inclusion
* Born at full term of pregnancy (≥ 37 weeks) with a birth weight ≥ 2.5 kg
* Informed consent form signed by one or both parents or by the legally acceptable representative and 1 or 2 independent witnesses
* Able to attend all scheduled visits and to comply with all trial procedures
* Has complied with the national immunization calendar (BCG for both countries) for the first 2 months of life.

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy
* Subjects with congenital or acquired immunodeficiency in the child's surrounding
* Systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion
* Blood or blood-derived products received since birth
* Any vaccination in the 4 weeks preceding the first trial vaccination
* Vaccination planned in the 4 weeks following the trial vaccination
* Documented history of pertussis, tetanus, diphtheria, poliomyelitis, Haemophilus influenzae type b or hepatitis B infection(s) (confirmed either clinically, serologically or microbiologically)
* Mother known as seropositive for HIV or Hepatitis C, or known carrier of Hepatitis B surface antigen
* Previous vaccination against pertussis, tetanus, diphtheria, poliomyelitis, or Haemophilus influenzae type b infection(s)
* Coagulopathy, thrombocytopenia or a bleeding disorder contraindicating IM vaccination
* History of seizures
* Febrile or acute illness on the day of inclusion.

Ages: 50 Days to 71 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2133 (Actual)
Dates: Start 2006-07; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Mexico City, Mexico
- Lima, Peru

REFERENCES:
- [Result] Macias M, Lanata CF, Zambrano B, Gil AI, Amemiya I, Mispireta M, Ecker L, Santos-Lima E. Safety and immunogenicity of an investigational fully liquid hexavalent DTaP-IPV-Hep B-PRP-T vaccine at two, four and six months of age compared with licensed vaccines in Latin America. Pediatr Infect Dis J. 2012 Aug;31(8):e126-32. doi: 10.1097/INF.0b013e318258400d. PMID 22531237
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated from 17 July 2006 to 02 January 2008 in 1 clinical center in Mexico and 1 clinical center in Peru.
Pre-assignment Details: A total of 2133 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- DTaP-IPV-Hep B-PRP~T: Participants received Diphtheria (D), tetanus (T), pertussis (acellular, component) (aP), hepatitis B (hep B [recombinant DNA]) and poliomyelitis (Inactivated [IPV]), and Haemophilus influenzae type b (Hib) conjugated vaccine adsorbed (DTaP-IPV-Hep B-PRP~T) plus a Placebo, oral poliovirus vaccine (OPV) in a 3-dose series with single doses at 2, 4, and 6 months of age.
- Tritanrix-Hep B/Hib™ + OPV: Participants received Tritanrix-Hep B/Hib™ + oral poliovirus vaccine (OPV) in a 3-dose series with single doses at 2, 4, and 6 months of age.
Period: Overall Study
Arm/Group | DTaP-IPV-Hep B-PRP~T | Tritanrix-Hep B/Hib™ + OPV
Started | 1422 (N for outcomes adjusted to include participant in Group 2 that got vaccine assigned to this group.) | 711 (A participant in this group mistakenly got Group 1 vaccine. N in outcomes adjusted accordingly.)
Completed | 1328 | 670
Not Completed | 94 | 41
Not completed — Serious adverse event | 6 | 1
Not completed — Adverse Event | 2 | 3
Not completed — Protocol Violation | 19 | 10
Not completed — Lost to Follow-up | 27 | 14
Not completed — Withdrawal by Subject | 39 | 12
Not completed — Did not meet age criteria | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTaP-IPV-Hep B-PRP~T | Tritanrix-Hep B/Hib™ + OPV | Total
Number analyzed (Participants) | 1422 | 711 | 2133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1422 | 711 | 2133
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months]
  Age Continuous | 1.89 (0.195) | 1.88 (0.197) | 1.88 (0.196)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 706 | 344 | 1050
  Male | 716 | 367 | 1083
Region of Enrollment [Number; unit: Participants]
  Mexico | 712 | 355 | 1067
  Peru | 710 | 356 | 1066

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With High Fever Observed After Either DTaP-IPV-Hep B-PRP~T or Tritanrix Hep B/Hib™ + Placebo or Tritanrix-Hep B/Hib™ + Placebo Injection.
Description: High fever was defined as rectal temperature equivalent to ≥ 39.6ºC.
Time Frame: Day 0 up to Day 7 post-injection
Population: The occurrence of high fever was assessed for all enrolled and vaccinated participants, intent-to-treat (safety) population. Total numbers of participants in each group adjusted for the participant that got a vaccine assigned for the other group.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP~T | Tritanrix-Hep B/Hib™ + OPV
Number analyzed (Participants) | 1423 | 710
Participants
  Post Any Dose (N = 1411, 703) | 56 | 39 [0 to 0]
  Post Dose 1 (N = 1408, 703) | 5 | 4 [0 to 0]
  Post Dose 2 (N = 1348, 681) | 25 | 15 [0 to 0]
  Post Dose 3 (N = 1328, 672) | 26 | 23 [0 to 0]

2. Secondary Outcome: Geometric Mean Titers of Anti Hepatitis B Antibodies Following Vaccination With Either DTaP-IPV-Hep B-PRP~T Vaccine + Placebo or Tritanrix-Hep B/Hib™ + Placebo
Description: Anti-hepatitis B (Hep B) antibodies were measured by automated enhanced chemiluminescence assay.
Time Frame: Day 30 post-dose 3
Population: Anti-hepatitis B antibody titers were assessed in a subset of the enrolled and vaccinated participants, intent-to-treat population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DTaP-IPV-Hep B-PRP~T | Tritanrix-Hep B/Hib™ + OPV
Number analyzed (Participants) | 184 | 95
Titers | 1075 [891 to 1298] | 3376 [2672 to 4338]

3. Secondary Outcome: Percentage of Participants Reaching Seroprotection Threshold Following Vaccination With Either DTaP-IPV-Hep B-PRP~T Vaccine + Placebo or Tritanrix-Hep B/Hib™ + Placebo
Description: Anti hepatitis B (Hep B) antibodies were measured by automated enhanced chemiluminescence assay.
  Two Seroprotection thresholds were defined: a titer ≥ 10 mIU/mL and ≥ 100 mIU/mL, respectively.
Time Frame: Day 30 post-dose 3
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | DTaP-IPV-Hep B-PRP~T | Tritanrix-Hep B/Hib™ + OPV
Number analyzed (Participants) | 184 | 95
Percentage of Participants
  ≥ 10 mIU/mL | 100 | 100 [0 to 0]
  ≥ 100 mIU/mL | 96 | 99 [0 to 0]

4. Secondary Outcome: Number of Participants Reporting at Least One Solicited Injection Site or Systemic Reaction Following Each Vaccination
Description: Solicited Injection Site Reactions: Pain, Erythema, Swelling. Solicited Systemic Reactions: Pyrexia (Temperature), Vomiting, Crying, Somnolence, Anorexia, Irritability.
  Severe solicited reactions were defined as follows: Pain, cries when injected limb is moved or the movement of the injected limb is reduced; Erythema and Swelling, ≥5 cm; Fever ≥39.6 ºC; Vomiting, ≥6 episodes per 24 hours or requiring parenteral hydration; Crying, >3 hours; Somnolence, sleeping most of the time or difficulty to wake up; Anorexia, refuses ≥3 feeds or refuses most feeds; Irritability, inconsolable.
Time Frame: Day 0 up to Day 7 Post-injection
Population: Solicited injection site and systemic reactions were assessed in the enrolled and vaccinated participants, intent-to-treat (safety) population. Total numbers of participants (N) in each group adjusted for the participant that got a vaccine assigned for the other group.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP~T | Tritanrix-Hep B/Hib™ + OPV
Number analyzed (Participants) | 1423 | 710
Participants
  Any Pain Post Dose 1 (N=1410, 703) | 831 | 574 [0 to 0]
  Severe Pain Post Dose 1 (N=1408, 703) | 175 | 193 [0 to 0]
  Any Pain Post Dose 2 (N=1348, 681) | 744 | 506 [0 to 0]
  Severe Pain Post Dose 2 (N=1348, 681) | 105 | 95 [0 to 0]
  Any Pain Post Dose 3 (N=1327, 672) | 519 | 448 [0 to 0]
  Severe Pain Post Dose 3 (N=1327, 672) | 29 | 65 [0 to 0]
  Any Erythema Post Dose 1 (N=1408, 703) | 245 | 234 [0 to 0]
  Severe Erythema Post Dose 1 (N=1408, 703) | 11 | 15 [0 to 0]
  Any Erythema Post Dose 2 (N=1348, 681) | 427 | 308 [0 to 0]
  Severe Erythema Post Dose 2 (N=1348, 681) | 6 | 16 [0 to 0]
  Any Erythema Post Dose 3 (N=1327, 672) | 587 | 340 [0 to 0]
  Severe Erythema Post Dose 3 (N=1327, 672) | 23 | 12 [0 to 0]
  Any Swelling Post Dose 1 (N=1406, 703) | 151 | 188 [0 to 0]
  Severe Swelling Post Dose 1 (N=1406, 703) | 8 | 24 [0 to 0]
  Any Swelling Post Dose 2 (N=1348, 681) | 259 | 270 [0 to 0]
  Severe Swelling Post Dose 2 (N=1348, 681) | 3 | 11 [0 to 0]
  Any Swelling Post Dose 3 (N=1327, 672) | 400 | 323 [0 to 0]
  Severe Swelling Post Dose 3 (N=1327, 672) | 3 | 7 [0 to 0]
  Any Pyrexia Post Dose 1 (N=1408, 703) | 538 | 473 [0 to 0]
  Severe Pyrexia Post Dose 1 (N=1408, 703) | 5 | 4 [0 to 0]
  Any Pyrexia Post Dose 2 (N=1348, 681) | 675 | 457 [0 to 0]
  Severe Pyrexia Post Dose 2 (N=1348, 681) | 27 | 16 [0 to 0]
  Any Pyrexia Post Dose 3 (N=1328, 672) | 552 | 445 [0 to 0]
  Severe Pyrexia Post Dose 3 (N=1328, 672) | 30 | 23 [0 to 0]
  Any Vomiting Post Dose 1 (N=1408, 703) | 230 | 120
  Severe Vomiting Post Dose 1 (N=1408, 703) | 10 | 4 [0 to 0]
  Any Vomiting Post Dose 2 (N=1348, 681) | 152 | 75 [0 to 0]
  Severe Vomiting Post Dose 2 (N=1348, 681) | 2 | 4 [0 to 0]
  Any Vomiting Post Dose 3 (N=1328, 672) | 167 | 95 [0 to 0]
  Severe Vomiting Post Dose 3 (N=1328, 672) | 17 | 10 [0 to 0]
  Any Crying Post Dose 1 (N=1409, 703) | 800 | 564 [0 to 0]
  Severe Crying Post Dose 1 (N=1409, 703) | 21 | 26 [0 to 0]
  Any Crying Post Dose 2 (N=1348, 681) | 721 | 481 [0 to 0]
  Severe Crying Post Dose 2 (N=1348, 681) | 9 | 8 [0 to 0]
  Any Crying Post Dose 3 (N=1327, 672) | 466 | 391 [0 to 0]
  Severe Crying Post Dose 3 (N=1327, 672) | 9 | 8 [0 to 0]
  Any Somnolence Post Dose 1 (N=1408, 703) | 635 | 375 [0 to 0]
  Severe Somnolence Post Dose 1 (N=1408, 703) | 46 | 26 [0 to 0]
  Any Somnolence Post Dose 2 (N=1348, 681) | 405 | 247 [0 to 0]
  Severe Somnolence Post Dose 2 (N=1348, 681) | 16 | 12 [0 to 0]
  Any Somnolence Post Dose 3 (N=1327, 672) | 272 | 204 [0 to 0]
  Severe Somnolence Post Dose 3 (N=1327, 672) | 12 | 11 [0 to 0]
  Any Anorexia Post Dose 1 (N=1408, 703) | 388 | 278 [0 to 0]
  Severe Anorexia Post Dose 1 (N=1408, 703) | 11 | 14 [0 to 0]
  Any Anorexia Post Dose 2 (N=1348, 681) | 327 | 195 [0 to 0]
  Severe Anorexia Post Dose 2 (N=1348, 681) | 12 | 11 [0 to 0]
  Any Anorexia Post Dose 3 (N=1327, 672) | 294 | 189 [0 to 0]
  Severe Anorexia Post Dose 3 (N=1327, 672) | 18 | 17 [0 to 0]
  Any Irritability Post Dose 1 (N=1408, 703) | 945 | 576 [0 to 0]
  Severe Irritability Post Dose 1 (N=1408, 703) | 42 | 47 [0 to 0]
  Any Irritability Post Dose 2 (N=1348, 681) | 799 | 492 [0 to 0]
  Severe Irritability Post Dose 2 (N=1348, 681) | 41 | 25 [0 to 0]
  Any Irritability Post Dose 3 (N=1327, 672) | 546 | 416 [0 to 0]
  Severe Irritability Post Dose 3 (N=1327, 672) | 11 | 17 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the day of the first injection (Day 0) through 6 months after the last injection.
Description: Total number of participants in each group adjusted for the participant that got a vaccine assigned for the other group. The number at risk for the solicited injection site and systemic reactions also reflects numbers with data.
Arm/Group | DTaP-IPV-Hep B-PRP~T | Tritanrix-Hep B/Hib™ + OPV
Serious Adverse Events (participants affected / at risk) | 91/1423 | 46/710
Other Adverse Events (participants affected / at risk) | 945/1423 | 576/710
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTaP-IPV-Hep B-PRP~T (N=1423) | Tritanrix-Hep B/Hib™ + OPV (N=710)
Cardio Respiratory Distress (Cardiac disorders) | 0 (0) | 1 (1)
Hip Dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Choledochal Cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess Neck (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 12 (12) | 6 (6)
Bronchopneumonia (Infections and infestations) | 13 (13) | 3 (3)
Encephalitis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 21 (21) | 18 (18)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 1 (1)
Kawasaki's disease (Infections and infestations) | 0 (0) | 1 (1)
Laryngotracheitis (Infections and infestations) | 2 (2) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Periorbital Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 3 (3)
Pneumonia viral (Infections and infestations) | 6 (6) | 2 (2)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Pyoderma (Infections and infestations) | 1 (1) | 0 (0)
Pyoderma Streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Encephalitis (Nervous system disorders) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1)
Febrile Convulsion (Nervous system disorders) | 4 (4) | 1 (1)
Hypotonic Hyporesponsive Episode (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Bronchial Hyperactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Foreign Body Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DTaP-IPV-Hep B-PRP~T (N=1423) | Tritanrix-Hep B/Hib™ + OPV (N=710)
Abdominal Pain (Gastrointestinal disorders) | 131/1411 (131) | 70/703 (70)
Diarrhoea (Gastrointestinal disorders) | 264/1411 (264) | 123/703 (123)
Solicited Vomiting Post-dose 1 (Gastrointestinal disorders) | 230/1410 (230) | 120/703 (120)
Solicited Injection site Erythema Post-dose 3 (General disorders) | 587/1410 (587) | 340/703 (340)
Injection Site Haemorrhage (General disorders) | 39/1411 (39) | 63/703 (63)
Injection Site Nodule (General disorders) | 81/1411 (81) | 79/703 (79)
Solicited Injection Site Pain Post-dose 1 (General disorders) | 831/1410 (831) | 574/703 (574)
Solicited Injection Site Swelling Post-dose 3 (General disorders) | 400/1408 (400) | 323/703 (323)
Solicited Irritability post-dose 1 (General disorders) | 945/1410 (945) | 576/703 (576)
Solicited Pyrexia Post-dose 2 (General disorders) | 675/1411 (675) | 457/703 (457)
Gastroenteritis (Infections and infestations) | 101/1411 (101) | 40/703 (40)
Nasopharyngitis (Infections and infestations) | 742/1411 (742) | 353/703 (353)
Pharyngitis (Infections and infestations) | 395/1411 (395) | 161/703 (161)
Rhinitis (Infections and infestations) | 136/1411 (136) | 56/703 (56)
Solicited Anorexia Post-dose 1 (Metabolism and nutrition disorders) | 388/1410 (388) | 278/703 (278)
Solicited Somnolence Post-dose 1 (Nervous system disorders) | 635/1410 (635) | 375/703 (375)
Solicited Crying Post-dose 1 (Psychiatric disorders) | 800/1411 (800) | 564/703 (564)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 163/1411 (163) | 74/703 (74)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 75/1411 (75) | 36/703 (36)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 160/1411 (160) | 54/703 (54)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.